CLINICAL TRIAL: NCT03579706
Title: Evaluation of a Brief, Online Intervention for Military Personnel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Norman Schmidt, Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Norr02
Record Dates: First submitted 2018-06-01; First posted 2018-07-06 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Experimental; Placebo Contol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants anonymously complete all online measures and the intervention without contact with study personnel. Participants are randomized to the active or control condition without being told which condition they are participating in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention condition will involve participants completing baseline measures, the Cognitive Anxiety Sensitivity Treatment, post measures, and a 4 month follow up assessment.
  Interventions: Behavioral: Cognitive Anxiety Sensitivity Treatment
- Control (Placebo Comparator): The control condition will involve participants completing baseline measures, the Physical Health Education Training, post measures, and a 4 month follow up assessment.
  Interventions: Behavioral: Physical Health Education Training

INTERVENTIONS:
Behavioral: Cognitive Anxiety Sensitivity Treatment — The Cognitive Anxiety Sensitivity Treatment is a computerized treatment that is a combination of psychoeducation plus interoceptive exposure for anxiety sensitivity (AS). The psychoeducational component will focus on the nature of stress and its effect on the body. Interoceptive exposure (IE) exercises, designed to correct the conditioned fear to these bodily sensations, will be explained and practiced.
  Arms: Intervention
Behavioral: Physical Health Education Training — The Physical Health Education Training is a computerized active placebo matched in time and structure to CAST that includes information about general health and wellness (e.g. diet, exercise etc.).
  Arms: Control

SUMMARY:
This randomized controlled trial will compare the effectiveness and acceptability of a computerized treatment targeting anxiety sensitivity compared to an active control: Physical Health Education Treatment (PHET) to determine efficacy among military personnel when delivered over the Internet.

Purpose: To investigate the efficacy and acceptability of a computerized stress sensitivity treatment delivered online among a population of U.S. military personnel.

DETAILED DESCRIPTION:
The objective of the current proposal is to evaluate the efficacy of the Cognitive Anxiety Sensitivity Treatment (CAST) program in an online RCT through Amazon's Mechanical Turk with Veterans and military personnel. The primary outcome variables will be traumatic stress, anxiety, and depressive symptoms. The study is being conducted at Florida State University.

Specific Aims: (1) Evaluate the efficacy of the CAST program delivered over the Internet among Veterans and military personnel; (2) Assess acceptability and usability of the CAST program delivered over the Internet without in person appointments; (3) Determine the feasibility of using Amazon's Mechanical Turk to recruit and conduct a fully online randomized controlled trial of a computerized treatment.

Veterans or active duty personnel (N = 100) who are at increased risk for mental health problems, as indicated by elevated anxiety sensitivity, will be recruited through Amazon's Mechanical Turk. Mechanical Turk is an online marketplace for individuals interested in completing computerized tasks, such as research surveys, for compensation. Participants will complete self-report symptom measures before and after the intervention as well as at a 4-month follow-up appointment. The intervention is a single session and lasts approximately 45 minutes. The intervention contains educational material to dispel commonly held false beliefs about the dangerousness of experiencing anxiety symptoms, for example elevated heart rate or a difficulty concentrating. Then participants are guided through an exercise designed to bring on these uncomfortable bodily sensations to help participants reduce the amount of distress these symptoms cause. Participants will also be asked to provide feedback related to acceptability and usability of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* current or past member of the U.S. military
* elevated anxiety sensitivity as indexed by ASI-3 cognitive concerns subscale

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Anxiety Sensitivity | Baseline; change from baseline to immediately post intervention, change from baseline to 4 month FU
  The Anxiety Sensitivity Index - 3 (ASI-3; Taylor et al., 2007) is an 18-item self-report measure of AS. This scale was developed to provide a more stable measure of the three most widely recognized AS subfactors (cognitive, social and physical concerns) than the original ASI provides. The measure has shown good psychometric properties (Taylor et al., 2007).

SECONDARY OUTCOMES:
Change in Anxiety Symptoms | Baseline; change from baseline to immediately post intervention, change from baseline to 4 month FU
  The Generalized Anxiety Disorder 7-item scale (GAD-7; Spitzer et al., 2006) is a 7- item self-report measure of generalized anxiety. Participants rate the frequency with which they experience anxiety-related symptoms on a scale of 0 (Not at all) to 3 (Nearly every day). The GAD-7 exhibited excellent internal consistency and good test-retest reliability (Spitzer et al., 2006). Total scores range from 0-21 with higher scores indicating greater anxiety symptoms.
Change in Depressive Symptoms Module (PHQ-9). | Baseline; change from baseline to immediately post intervention, change from baseline to 4 month FU
  The Patient Health Questionnaire - Depression (PHQ-9) is the 9-item depression module of the larger Patient Health Questionnaire (PHQ;Spitzer et al., 1999) which was designed to assess eight DSM-IV diagnoses, including major depressive disorder. The PHQ-9 exhibited excellent internal reliability and excellent test-retest reliability (Kroenke et al., 2001). Total scores range from 0-27 with higher scores indicating greater depressive symptoms.
Change in Post-Traumatic Stress Disorder Symptoms | Baseline; change from baseline to immediately post intervention, change from baseline to 4 month FU
  The Post-Traumatic Stress Disorder Checklist for DSM-5 (PCL-5) is a brief, 20-item self-report instrument that assesses the 20 DSM-5 symptoms of posttraumatic stress disorder. We will use the PCL-5 to obtain total symptom severity scores and DSM-5 symptom cluster severity scores for each participant.
Usability of the computerized intervention | Immediately post intervention
  The System Usability Scale (SUS) is a 10 item self-report questionnaire assessing general usability of a given program (Brooke, 1996). The SUS total score ranges from 5 to 50 with higher scores indicating better usability.
Client Satisfaction | Immediately post intervention
  The Client Satisfaction Questionnaire (CSQ) is an 8 item self-report questionnaire assessing general satisfaction with services of treatment received by the individual (Attkisson and Zwick, 1982). The CSQ has shown high reliability and internal consistency (Attkisson and Zwick, 1982). Total score ranges from 8 to 32 with higher scores indicating greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Norman B Schmidt, PhD, Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No